CLINICAL TRIAL: NCT03460275
Title: Osimertinib as First-line Therapy for Patients With EGFR Mutation-positive Locally Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer(NSCLC), a Single-Arm, Open-Lable, Prospective, Multicenter, Phase II Clinical Trial
Brief Title: Osimertinib as First-line Therapy for Patients With Late-stage Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hao Long, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2018-001
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Other): Osimertinib Mesylate Tablets 80 mg, one time a day until disease progression
  Interventions: Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: Osimertinib Mesylate Tablets — Osimertinib 80mg oral administration daily until progression or occurring intolerable treatment-related toxic effects or patients withdrawing informed consent(Based on whichever occurs first)

SUMMARY:
Based on the existing research results, Osimertinibi is effective not only for patients with sensitizing EGFR mutations, but also for other less common EGFR mutations. However, no studies have been done so far regarding the difference in efficacy of various EGFR mutation subtypes. Meanwhile, the presenting studies data of the safety and efficacy of Osimertinib as first-line therapy for NSCLC is very limited. Therefore, this study aims at assessing the safety and efficacy of Osimertinib as First-line therapy for patients with EGFR mutation-positive locally advanced or Metastatic Non-squamous NSCLC as well as the its difference in efficacy of various EGFR mutation subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable locally advanced(Stage IIIB，not amenable to definitive multi-modality therapy)、metastatic(Stage IV)or recurrent EGFR mutation-positive Non-squamous NSCLC.( Diagnosis of NSCLC based on sputum cytology alone is not acceptable; If the specimen shows more than one tumor components, a pathological evaluation to classify the major histological subtype of the lung cancer must be performed.)Choose EGFR-TKIs as the first-line therapy.
2. Patients with EGFR mutation(any form of EGFR mutation subtype except for EGFR exon 20 insertion mutation) detected by First generation sequencing(Sager sequencing) or next generation sequencing(NGS) from tissue sample includes fresh tissue or formalin-fixed paraffin-embedded(FFPE)sample or body fluid sample(blood, pleural effusion, cerebrospinal fluid ,etc.)
3. Measurable disease by RECIST 1.1(At least one lesion that can be accurately measured at baseline as ≥10mm in the longest diameter, If the CT scan thickness >5mm, the lesion diameter is at least 2 times the scan thickness).
4. Age≥18 years or≤75 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)of 0 or 1.
6. Estimated survival time(EST) no less than 12 weeks.
7. Adequate hematologic function:Absolute neutrophil count(ANC) ≥1.2 x 10^9/L;Platelets≥100 x 10^9/L;Hemoglobin≥9 g/dL(can be maintained by blood transfusion and exceeding 9 g/dL).
8. Adequate hepatic function:Total bilirubin < 1.5 x upper limit of normal(ULN);For patients without liver metastases:Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) <2.5 x ULN;For patients with known hepatic metastases AST and ALT both <5 x ULN.
9. Adequate renal function:Serum Creatinine≤1.5x ULN or creatinine clearance≥50mL/min;
10. Within 7 days before included in the study:International normalized ratio(INR) ≤1.5, prothrombin time(PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
11. Patients is willing and able to comply with the protocol for the duration of the study including scheduled visits and examinations including following up.
12. Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

1. Pathologic evaluation indicates NSCLC mixes with small-cell lung cancer(SCLC), adenosquamous carcinoma with component of squamous cell carcinoma comprises major part of the tumor.
2. Prior therapy with 1)EGFR-TKIs such as Erlotinib and Gefitinib;2)EGFR inhibitor such as Cetuximab.
3. Prior treatment with any systemic anti-cancer therapy for NSCLC including cytotoxic chemotherapy, targeted therapies(such as monoclonal antibody like Trastuzumab), investigational treatment(Do not include previously received adjuvant therapy or neoadjuvant therapy(adjuvant chemotherapy/radiation therapy(RT)).
4. Radiotherapy treatment with a wide field of radiation for bone metastases to more than 30% of the bone marrow within 4 weeks of study entry; major surgery(including open surgical biopsy within 4 weeks prior to the administration of the study drug; Suffer major injuries; planned major surgery during the study.
5. Patients with Spinal cord compression, severe neurological symptoms and unstable brain metastases (except for those patients who are asymptomatic or have had a stable neurological status for at least 2 weeks after symptomatic or supportive therapy).
6. Patients currently receiving medications or herbal supplements known to be potent inducers of cytochrome P450 or potent inhibitors or inducers of CYP3A4.
7. Physiological malfunction of upper digestive tract; malabsorption syndrome; Inability to swallow the formulated product.
8. Any clinical evidence indicates:1) moderate to severe chronic obstructive pulmonary disease (COPD)[history of COPD or exposure to high risk factor for the disease; pulmonary function tests: forced expiratory volume in one second(FEV1)<80 %predicted, FEV1/ FVC<70%;With/without symptoms: shortness of breath, chronic cough, sputum production] ; 2)active interstitial lung disease(ILD)[ pulmonary function tests: FEV1/ FVC<70%, FEV1<80 %predicted, diffusing capacity of the lung for carbon monoxide (DLCO)< 40%;high-resolution computed tomography(HRCT) confirmed diffuse pulmonary interstitial lesions].
9. Any diseases, metabolic disorders, physical examinations or laboratory results indicate the patient may have contradictions of the study drug or high risk factors of treatment-related complications.
10. Any evidence of severe or uncontrolled systemic diseases, including active infection;uncontrolled hypertension;unstable angina; Angina within 3 months prior to study; congestive heart failure (NYHA Grade II or greater); prior myocardial infarction (NSTEMI or STEMI) within 6 months prior to study enrollment; severe arrhythmia requiring medical treatment; hepatic, renal or metabolic diseases.
11. Active infection of human immunodeficiency virus (HIV).
12. Patients with unhealing wound ,active peptic ulcer or bone fracture.
13. Females who are 1)pregnant;2)breastfeeding;3)of reproductive potential planning to become pregnant; Males and females who are not using an effective method of birth control.
14. History of allergic reactions attributed to compounds, or any of its excipients, of similar chemical or biologic composition to Osimertinib.
15. Judgment by the Investigator that the patient should not participate in the study if the conditions of the patient is likely to compromise the efficacy and safety of the study or if the patient is unlikely to comply with study procedures, restrictions and requirements.
16. Malignancies except for NSCLC requiring treatments within the past 2 years prior to the administration of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 | eight weeks
  Patients were images with computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat sen University cancer center, Guangzhou, Guangdong